CLINICAL TRIAL: NCT05449912
Title: ENVI-MI (Environment and Myocardial Infarction) : Impact of Environmental Exposure at Home Address on One-year Post-myocardial Infarction Survival
Brief Title: Impact of Environmental Exposure at Home Address on One-year Post-myocardial Infarction Survival
Acronym: ENVI-MI
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Other Study IDs: Cottin Fondation Cœur 2018
Record Dates: First submitted 2022-07-05; First posted 2022-07-08 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Myocardial Infarction
MeSH Terms: conditions — Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients registered in the RICO database: Patients hospitalized for myocardial infarction between 01/01/2002 and 31/12/2008
  Interventions: Other: Collection of environmental exposure data

INTERVENTIONS:
Other: Collection of environmental exposure data — noise pollution air pollution proximity and accessibility to green spaces, blue spaces

SUMMARY:
Numerous studies have explored the effects of environmental exposure to noise, air pollution and proximity to "natural" areas on various conditions. However, very few studies have focused on the "post-diagnosis" follow-up of patients after hospitalization for an ischemic cardiovascular episode and, to our knowledge, none have examined patient evolution at one year after myocardial infarction. Thus, the real influence of factors and pollutants widely represented in the urban environment, in particular air pollution, noise pollution, and proximity and accessibility to natural areas ("green" or "blue" spaces), on the evolution of post-myocardial infarction at one year remains to be identified and quantified.

The objective of the ENVI-MI project is to evaluate the impact of environmental exposure in the place of residence (noise, air pollution, proximity to "natural" spaces) on the evolution of post-myocardial infarction at one year within the Dijon metropolitan area.

ELIGIBILITY:
Inclusion Criteria:

Patient :

* registered in the RICO database
* hospitalized for MI between January 1, 2002 and December 31, 2008,
* whom residence is located in one of the 15 communes of the Dijon urban unit (except for patients living in the area subject to the noise exposure plan of the military airport)

Exclusion Criteria: NA

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients registered in the RICO database
Sampling Method: Non-Probability Sample
Enrollment: 982 (Actual)
Dates: Start 2019-02-18 (Actual); Primary Completion 2020-02-28 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Occurrence of a cardiovascular event | 1 year
  Occurrence of any of the following cardiovascular events during the 1-year follow-up: death, recurrence, or rehospitalization for CV causes

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Dijon Bourogne, Dijon, France

REFERENCES:
- [Result] Koczorowski M, Bernard N, Mauny F, Chague F, Pujol S, Maza M, Cottin Y, Zeller M; ENVI-MI Study Group. Environmental noise exposure is associated with atherothrombotic risk. Sci Rep. 2022 Feb 24;12(1):3151. doi: 10.1038/s41598-022-06825-0. PMID 35210480